CLINICAL TRIAL: NCT00111917
Title: Clinical Efficacy of Remicade in Chronic Beryllium Disease: A Randomized, Double-Blind, Placebo-Controlled, Investigator Initiated Trial
Brief Title: Beryllium Infliximab Study: Clinical Interventional Trial
Acronym: BISCIT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not enough patients meeting criteria to enroll in the time period
Sponsor: Maier, Lisa, M.D. (Individual)
Collaborators: Centocor, Inc. (Industry); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NJ202; 1UL1RR025780 (NIH)
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-03

CONDITIONS: Berylliosis; Beryllium Disease
Keywords: Chronic Beryllium Disease; Berylliosis; Beryllium Disease; CBD; Infliximab
MeSH Terms: conditions — Berylliosis | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab (Experimental): infusion: 3:1 infliximab:placebo ratio administered at 0, 2, 6, 12, 18 and 24 weeks.
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): infusion: 3:1 infliximab:placebo ratio administered at 0, 2, 6, 12, 18 and 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Infliximab — anti-TNF
  Other Names: Remicade
  Arms: Infliximab
Other: Placebo — Placebo infusion
  Arms: Placebo

SUMMARY:
The goal of this research study is to test the clinical effectiveness of a drug called infliximab (Remicade) in chronic beryllium disease (CBD). This drug may reduce tumor necrosis factor-alpha (TNF-a), which is associated with more severe disease and inflammation in the lung. Receiving infliximab may help with symptoms, and may improve clinical testing data normally ordered by your doctor, such as breathing tests. Baseline and follow-up testing will look for improvements in breathing tests (pulmonary function testing), exchange of oxygen in the lungs (exercise test), chest x ray, and lung inflammation.

DETAILED DESCRIPTION:
Hypothesis:

The central hypothesis of this study is that infliximab will prove to be efficacious in the treatment of chronic beryllium disease (CBD), and that it will do so by inhibiting beryllium specific T cell proliferation and cytokine production.

Specific Aims:

Specific Aim 1: To determine the clinical effectiveness of infliximab on chronic beryllium disease. The efficacy of infliximab will be measured by improvement in arterial gas exchange, or arterial alveolar oxygen gradient (A-ad02) at end exercise in subjects with CBD who remain symptomatic and with pulmonary impairment despite current treatment with prednisone and/or methotrexate. Secondary outcome measures will include change in airflow, lung volume, diffusing capacity (DLCO), profusion of small opacities on chest x-ray, dyspnea score, and quality of life questionnaires.

Specific Aim 2: To determine the effect of infliximab on intermediate markers of biological function in CBD. In vitro studies will examine the effect of infliximab on blood and lung cells in culture, as measured by a decrease in beryllium (Be)-stimulated lymphocyte proliferation; a decrease in Be-stimulated cytokine production, including TNF-a, IFN-g, and IL-2; altered Be-stimulated apoptosis of macrophages or lymphocytes.

Research Design and Methods: Since no information is available regarding the pharmacokinetics of infliximab in patients with CBD, the pharmacokinetic information available from the use of infliximab in other similar inflammatory conditions formed the basis for selecting the dose regimen for this protocol. Particularly, a 5mg/kg dose will be used for this study, based on the dose selection used in the sarcoidosis protocol C0168T48 presently underway in a multi-center trial (NJC IRB HS-1771).

This is an investigator initiated, 40 week, randomized, double-blind, placebo controlled study to evaluate the efficacy of infliximab dosed at 5mg/kg, compared to placebo, in individuals with symptomatic CBD with pulmonary involvement despite prednisone and/or methotrexate treatment. Infliximab or placebo will be infused at weeks 0, 2, 6, 12, 18, and 24 including spirometry, lung volumes and DLCO. Approximately 20 participants will be enrolled in the study at National Jewish Medical and Research Center at a 3:1 drug: placebo rate.

The primary endpoint of this study will be a change from baseline testing to week 28 testing in the A-adO2 at end exercise on a 6 minute walk. At baseline evaluation, subjects will undergo full pulmonary function testing, a blood draw for the beryllium lymphocyte proliferation test (BeLPT), 6 minute walk, chest x-ray, and quality of life and dyspnea questionnaires. Follow-up full pulmonary function testing, rest and end exercise A-ad02, pulse oximetry with total distance (workload) achieved on a 6 minute walk, and chest radiograph will be measured at week 12. Final outcome measurements (same as baseline testing), including bronchoscopy with BAL, will be repeated at week 28. A follow-up appointment will be scheduled at week 40 to assess patients' general health, as well as measure rest and end exercise A-ad02 and pulse oximetry with 6 minute walk, pulmonary function test, QOL/dyspnea scoring, and chest radiograph interstitial lung opacity profusion score.

The effects of infliximab on the Be-stimulated immune response will be assessed by comparing the following markers before and after infliximab therapy: 1. BeLPT from blood and lavage cells (BAL); 2. Be-stimulated cytokine production from BAL cells including TNF-a, IFN-γ, and IL-2; 3. Cell-specific apoptosis. The assay will include an unstimulated control, 100 mM BeSO4, 100 mM Al2(SO4)3 metal-salt control, PHA - lymphocyte proliferation control, infliximab control, infliximab + BeSO4, infliximab + Al2(SO4)3. At days 4, 5, and 6 after Be exposure, the wells are pulsed with the DNA-specific precursor, 3H-TdR, incubated for four hours, harvested on glass fiber filters, and liquid scintillation methods are used for counting. Results are reported as a stimulation index, which is a ratio of the counts per minute of the treatment group to the counts per minute of the unstimulated group. To determine the effect of infliximab on cytokine production, CBD BAL and CBD PBMC will be stimulated with Be for 24 hours. ELISA will be used to determine TNF-α, IFN-γ, and IL-2 supernatant levels. After 24 hours of beryllium exposure, we will harvest supernatants and perform ELISA testing for TNF-α, IFN-γ, and IL-2. In order to determine if infliximab causes an increase in lymphocyte or macrophage apoptosis, CBD BAL cells will be cultured for 24 hours with Be. Cells will be double stained for CD4+ (Th1) and CD71+ macrophages versus intracellular activated caspase-3, caspase-8 and caspase-9. These in vitro studies will be used to assess the potential biologic function of infliximab on immune mediated diseases using a disease model with known antigen, CBD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-80.
* Noncaseating granulomas and/or mononuclear cell infiltrates demonstrated on transbronchial lung biopsy.
* Abnormal blood and/or BAL BeLPT results.
* Current treatment with prednisone and/or methotrexate specifically for CBD and not any other condition, at any range of dosage, for at least 6 months prior to enrollment, and on a stable dosage for at least 1 month prior to first infusion.
* Moderate CBD severity, such that participants can safely undergo bronchoscopy with BAL including PaO2 >= 50 mmHg on room air (at Denver altitude of 5,280 ft).
* Availability to come back to National Jewish Medical and Research Center for infusions, evaluations, and follow-ups.
* Capable of providing informed consent.
* Willing and able to adhere to the study visit schedule and other protocol-specified procedures.

Exclusion Criteria:

* Positive tuberculosis (TB) skin test upon screening: An intradermal tuberculin skin test must be performed within 1 month prior to the first administration of study agent.
* Any evidence of TB.
* Considered ineligible according to the TB eligibility assessment, screening, and early detection of reactivation rules.
* Positive pregnancy test.
* Women who are pregnant, nursing, or planning pregnancy within one year after screening
* Contraindications to bronchoscopy and BAL such as bleeding diathesis, PaO2 <50 mmHg on room air, evidence of acute infection, hemodynamic instability with labile blood pressure, either <90/60 or >160/110, untreated coronary artery disease, or other medical reason for which a subject will not be able to safely undergo bronchoscopy.
* Positive cultures from prior BAL indicating mycobacterial or fungal infection.
* Positive special stains for acid fast bacilli (AFB) or fungi on prior lung biopsies.
* Known atypical mycobacterium infection.
* Clinical evidence of active infection at time of enrollment.
* Serious acute infections (e.g., viral hepatitis, pneumonia or pyelonephritis) in the previous 3 months.
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Documented HIV infection.
* Positive serology for active hepatitis B or C. A positive result will indicate the need for referral to a consultant Hepatologist for further investigation and support.
* Use of any investigational drug within 1 month prior to screening or within 5 half lives of the investigational agent, whichever is longer.
* Treatment with any other therapeutic agent targeted at reducing TNF-a (e.g. pentoxifylline, thalidomide, etanercept, etc.) within 3 months of screening.
* Prior use of Enbrel® or Humera®.
* Previous administration of infliximab.
* Known allergy to murine (mouse) products.
* Have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis).
* Any history of congestive heart failure, severe right sided heart failure, or cor pulmonale.
* Presence of a transplanted organ (with the exception of a corneal transplant > 3 months prior to screening).
* Major surgery in the previous 3 months.
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* History of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or perioaortic areas), or splenomegaly.
* Known recent substance abuse (drug or alcohol).
* Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Maier, MD,MSPH, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Maier LA, Barkes BQ, Mroz M, Rossman MD, Barnard J, Gillespie M, Martin A, Mack DG, Silveira L, Sawyer RT, Newman LS, Fontenot AP. Infliximab therapy modulates an antigen-specific immune response in chronic beryllium disease. Respir Med. 2012 Dec;106(12):1810-3. doi: 10.1016/j.rmed.2012.08.014. Epub 2012 Sep 11. No abstract available. PMID 22974830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We aimed to enroll 20 CBD subjects on stable doses of corticosteroids and/or methotrexate, with no evidence of active or chronic infection, malignancy, other chronic disease, or past treatment with another biologic with a 3:1 infliximab:placebo ratio
Pre-assignment Details: the sponsor stopped the study due to slow recruitment
Groups:
- Group 1 - Infliximab: This group was given an infusion of inliximab
- Group 2 - Placebo: This group was given a placebo infusion
Period: Overall Study
Arm/Group | Group 1 - Infliximab | Group 2 - Placebo
Started | 9 | 4
Completed | 8 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Infliximab: patients who will be placed on infliximab and controls who will get placebo
- Control: CBD placed on placebo
- Total: Total of all reporting groups
Arm/Group | Infliximab | Control | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Continuous [Mean (Full Range); unit: years] — patient reported age
  years | 54.63 [46 to 65] | 69.75 [67 to 74] | 56.5 [46 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Post Hoc Outcome: Absolute Numbers of Lymphocytes
Description: Absolute number of lymphocytes*10^6/cc in blood
Time Frame: after 28 week follow-up
Measure: Median (Standard Error); unit: absolute number*10^6/cc
Groups:
- Infliximab: Infliximab infusion
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 8 | 2
absolute number*10^6/cc | 1.7 (0.18) | 1.02 (0.56)

2. Primary Outcome: A-a Gradient at End Exercise
Description: change in end-exercise A-a gradient
Time Frame: after 28 week follow-up. The Alveolar-arterial gradient (A-a gradient), is a measure of the difference between the alveolar partial pressure (A) of oxygen and the arterial (a) partial pressure of oxygen
Population: Accurate measures were not obtained on all patients at both timepoints.
Measure: Median (Standard Error); unit: mmHg
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 7 | 2
mmHg | 27.3 (10.56) | 94.17 (18.73)

3. Post Hoc Outcome: BAL WBC/cc
Description: WBC * 10^6/cc in bronchalveolar lavage
Time Frame: after 28 weeks
Measure: Median (Standard Deviation); unit: absolute WBC*10^6/cc
Groups:
- Infliximab: Infliximab received
- Placebo: Placebo received
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 5 | 2
absolute WBC*10^6/cc | 0.23 (0.04) | 0.25 (0.03)

4. Post Hoc Outcome: BAL % Lymphocytes
Description: % of WBCs that are lymphocytes in bronchoalveolar lavage
Time Frame: after 28 week infusion
Measure: Median (Standard Deviation); unit: percentage of lymphocytes in BAL
Groups:
- Group 1: Infliximab
- Group 2: Placebo received
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 5 | 2
percentage of lymphocytes in BAL | 4.68 (7.84) | 14.7 (0)

ADVERSE EVENTS:
Time Frame: through week 40
Description: adverse events reported through week 40
Groups:
- Group 1 - Infliximab: Infliximab infusion received
- Group 2 - Placebo: Placebo infusion received
Arm/Group | Group 1 - Infliximab | Group 2 - Placebo
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Infliximab (N=8) | Group 2 - Placebo (N=3)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Nausea, vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
liver function levels (Hepatobiliary disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Although our goal was 20 CBD subjects, only 11 subjects were enrolled, 8:3 in the infliximab:placebo treatment arms as the study was stopped by the sponsor due to slow recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No